CLINICAL TRIAL: NCT00973024
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Dose-Loading Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42160443 as Adjunctive Therapy in Subjects With Inadequately Controlled, Moderate to Severe, Chronic Low Back Pain
Brief Title: A Dose-ranging Study of the Safety and Effectiveness of JNJ-42160443 as add-on Treatment in Patients With Low Back Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on lack of efficacy in PAI2003, sponsor made the decision to discontinue the trial.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016468; 42160443PAI2003 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2009-009857-17 (EudraCT Number)
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain; Low Back Pain, Recurrent
Keywords: JNJ-42160443; Low back pain-related pain; moderate to severe, chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- JNJ-42160443 1 mg (Experimental)
  Interventions: Drug: JNJ-42160443 1 mg; Drug: Matching Placebo
- JNJ-42160443 3 mg (Experimental)
  Interventions: Drug: JNJ-42160443 3 mg; Drug: Matching Placebo
- JNJ-42160443 6 mg/3mg (Experimental)
  Interventions: Drug: JNJ-42160443 6 mg/3mg; Drug: Matching Placebo
- JNJ-42160443 10 mg (Experimental)
  Interventions: Drug: JNJ-42160443 10 mg; Drug: Matching Placebo

INTERVENTIONS:
Drug: JNJ-42160443 3 mg — JNJ-42160443: type=exact number, unit=mg, number= 3, form=solution for injection, route=Subcutaneous use or Placebo: form=solution for injection, route=Subcutaneous injection. One inj of 3 mg of JNJ-42160443 or matching placebo every 4 wks for up to 104 wks.
  Arms: JNJ-42160443 3 mg
Drug: JNJ-42160443 1 mg — JNJ-42160443: type=exact number, unit=mg, number= 1, form=solution for injection, route=Subcutaneous use or Placebo: form=solution for injection, route=Subcutaneous injection. One inj of 1 mg of JNJ-42160443 or matching placebo every 4 wks for up to 104 wks.
  Arms: JNJ-42160443 1 mg
Drug: JNJ-42160443 6 mg/3mg — JNJ-42160443: type= exact number, unit= mg, number= 3 and 6, form=solution for injection, route= Subcutaneous use or Placebo: form= solution for injection, route= Subcutaneous injection. 1 inj of 6 mg of JNJ-42160443 on Day 1 followed by 1 inj of 3 mg or matching placebo every 4 wks for up to 104 wks.
  Arms: JNJ-42160443 6 mg/3mg
Drug: JNJ-42160443 10 mg — JNJ-42160443 10 mg: type=exact number, unit=mg, number= 10, form=solution for injection, route=Subcutaneous use or Placebo: form=solution for injection, route=Subcutaneous injection. One inj of 10 mg of JNJ-42160443 or matching placebo every 4 wks for up to 104 wks.
  Arms: JNJ-42160443 10 mg
Drug: Matching Placebo — Form= solution for injection, route= subcutaneous. Matching placebo given as a subcutaneous (SC) (under the skin) injection (inj) once every 4 weeks (wks).

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of different doses of JNJ-42160443 with placebo in the treatment of chronic, moderate to severe low back pain patients with a diagnosis of chronic low back pain.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the physician nor the patient knows the name of the assigned drug) study to evaluate the safety and effectiveness of different doses of JNJ-42160443 compared with placebo in the treatment of patients with a diagnosis of chronic low back pain who have moderate to severe, chronic low back pain that is not controlled by standard pain medications. JNJ-42160443 (10 mg/ml) or matching placebo given as a subcutaneous (SC) (under the skin) injection (inj) once every 4 weeks (wks); one of four JNJ-42160443 doses (1 mg every 4 wks; 3 mg every 4 wks; 6 mg loading dose on Day 1 followed by 3 mg every 4 wks; or 10 mg every 4 wks, or matching placebo for up to 104 wks (12-wk double-blind efficacy period + 92-wk double-blind extension period).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic low back pain

Exclusion Criteria:

* Pain with radiation to the extremity and with neurologic signs
* history within the past year of any of the following: seizure disorder
* intrathecal therapy and ventricular shunts, mild or moderate traumatic brain injury, stroke, or transient ischemic attack, meningitis
* History of brain injury within the past 15 years consisting of >= 1 of the following, or with residual sequalae suggesting transient changes in consciousness: brain contusion, intracranial hematoma, either unconsciousness or posttraumatic amnesia lasting more than 24 hours
* History of epilepsy or multiple sclerosis
* Current diagnosis of fibromyalgia, complex regional pain syndrome (including reflex sympathetic dystrophy or causalgia), acute spinal cord compression, bowel or bladder dysfunction as a result of cauda equine compression, back pain caused by secondary infection, or pain caused by confirmed or suspected neoplasm
* Any new or unresolved neurologic deficits, including progressive deficits, within 6 months before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average low back pain-related pain intensity score | At the end of the 12-week double-blind efficacy phase

SECONDARY OUTCOMES:
Change from baseline in the ODI subscale and total scores | At the end of the 12-week double-blind efficacy phase
Change from baseline in the pain severity and pain interference subscales of the BPI Short Form | At the end of the 12-week double-blind efficacy phase
Changes in PGA scores | At the end of the 12-week double-blind efficacy phase
Change from baseline in the pain severity and pain interference subscales of the Brief Pain Inventory (BPI) Short Form | At the end of the 12-week double-blind efficacy phase
Changes in Patient Global Assessment (PGA) scores | At the end of the 12-week double-blind efficacy phase
Change from baseline in the Oswestry Disability Index (ODI) subscale and total scores | At the end of the 12-week double-blind efficacy phase

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (60):
- United States (41):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Pismo Beach, California
  - San Diego, California
  - Hollywood, Florida
  - Oldsmar, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Eagle, Idaho
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Valparaiso, Indiana
  - West Des Moines, Iowa
  - Prairie Village, Kansas
  - Topeka, Kansas
  - Baton Rouge, Louisiana
  - Lake Charles, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Watertown, Massachusetts
  - East Lansing, Michigan
  - Williamsville, New York
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington
- Belgium (3):
  - Edegem
  - Genk
  - Leuven
- Canada (15):
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Greater Sudbury, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec
- Maastricht, Netherlands

REFERENCES:
- [Derived] Sanga P, Polverejan E, Wang S, Kelly KM, Thipphawong J. Efficacy, Safety, and Tolerability of Fulranumab as an Adjunctive Therapy in Patients With Inadequately Controlled, Moderate-to-Severe Chronic Low Back Pain: A Randomized, Double-blind, Placebo-controlled, Dose-ranging, Dose-loading Phase II Study. Clin Ther. 2016 Jun;38(6):1435-1450. doi: 10.1016/j.clinthera.2016.03.030. Epub 2016 Apr 18. PMID 27101815